CLINICAL TRIAL: NCT00262639
Title: A Double Blind Evaluation of Flumazenil and Gabapentin for the Treatment of Alcohol Withdrawal and Relapse Prevention
Brief Title: Prometa Protocol for Alcohol Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Raymond F. Anton, Distinguished University Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15844
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Results first posted 2009-08-14 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Alcohol Dependence
Keywords: Alcoholism; Alcohol Dependence; Alcohol Withdrawal; Treatment; Pharmacotherapy
MeSH Terms: conditions — Alcoholism | interventions — Flumazenil; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): 2 mg flumazenil given over 20 minutes on Day 1 and Day 2. Gabapentin 300 mg Day 1; gabapentin 600 mg Day 2; gabapentin 900 mg Day 3; gabapentin 1200 mg Day 4 to 30; gabapentin 900 mg day 31-33; gabapentin 600 mg day 34-36; gabapentin 300 mg day 37-39.
  Interventions: Drug: Flumazenil and Gabapentin
- II (Placebo Comparator): 20 mg Saline infused slowly over 20 minutes. Placebo 1 capsule Day 1, 2 capsules Day 2, 3 capsules Day 3, 4 capsules days 4 to 30; 3 capsules Day 31 to 33; 2 capsules day 34 to 36 and 1 capsule 37 to 39.
  Interventions: Drug: Flumazenil and Gabapentin; Drug: Placebo

INTERVENTIONS:
Drug: Flumazenil and Gabapentin — 2 mg flumazenil for infusion given slowly over 20 minutes given day 1 and day 2 gabapentin 300 mg increasing to 1200 mg over 4 days and continuing to day 30. Gabapentin 900 mg Day 31 to Day 33 gabapentin 600 mg Day 34 to 36 and gabapentin 300 mg Day 37 to 39.
Drug: Placebo — 20 mg Saline infused slowly over 20 minutes. Placebo 1 capsule Day 1, 2 capsules Day 2, 3 capsules Day 3, 4 capsules days 4 to 30; 3 capsules Day 31 to 33; 2 capsules day 34 to 36 and 1 capsule 37 to 39.
  Arms: II

SUMMARY:
This is a placebo controlled trial (some people receive active and some people receive inactive medication) to evaluate the effectiveness of a new protocol to treat alcohol dependence. Two main medications (plus ancillary non-placebo controlled medications) and their placebos (inactive drugs) will be utilized to treat both alcohol withdrawal, promote abstinence, and reduce drinking over approximately a six-week treatment period. All participants will meet criteria for Alcohol Dependence and be drinking heavily up until 72 hours prior to receiving the first study drug. They will be injected one drug (flumazenil or placebo) over a two day period and receive the second one (gabapentin or placebo) by mouth for 39 days. The main hypothesis is that this protocol will reduce early alcohol withdrawal symptoms and will reduce relapse to drinking and promote abstinence compared to the placebo (inactive) drug group. Secondary outcomes that will be evaluated include reduction in craving, improvement in sleep, brain activity and mood.

DETAILED DESCRIPTION:
Approximately 60 alcohol dependent individuals who are drinking heavily up until 72 hours, or less, prior to study participation will be randomized to receive either flumazenil (intravenously)on two successive days and gabapentin (orally)for 39 days or their matching placebos. They also will receive hydroxyzine and vitamins. Individuals will be evaluated for alcohol withdrawal, their response to acoustic startle, cognitive ability, craving, mood, sleep and drinking during the first week. They will then be seen weekly for about 6 weeks during which they take gabapentin or placebo and are provided with Combined Behavioral Intervention Therapy (counseling) once a week, or more, as required. Over this period they will be evaluated weekly for alcohol consumption, craving, sleep, mood, and biological markers of alcohol consumption ( percent carbohydrate deficient transferrin and gamma-glutamyl transferase). Blood will be obtained on week 3 and 6 for general health (liver, blood count etc.) screening. After the end of treatment, subjects will be followed-up at 4 weeks and again at 8 weeks after treatment to evaluate alcohol consumption, craving, sleep, mood.

Subjects will undergo a functional magnetic resonance imaging (MRI) procedure sometime during the second or third week of study medication to assess cue induced regional brain activation to investigate the effect of medication on brain response to alcohol visual cues.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 70.
2. Participants will meet criteria for primary DSM IV alcohol dependence, drink on at least 70% of days in the last 30 days prior to assessment, and drink at least 5 drinks per drinking day.
3. No more than 72 hours since last drink of alcohol. Rationale: to focus on symptoms occurring during the early alcohol cessation period.
4. Low CIWA-Ar group: have a CIWA-Ar score less than or equal to 6; High CIWA-Ar group: have a CIWA-Ar score greater than or equal to 7 but less than or equal to 15.
5. Able to read and understand questionnaires and informed consent.
6. Has stable housing for past 3 months.

Exclusion Criteria:

1. Currently meets DSM-IV criteria for any other psychoactive substance dependence disorder except nicotine dependence.
2. Any psychoactive substance abuse, except marijuana and nicotine, within the last 30 days as evidenced by subject report or urine drug screen.
3. Meets DSM-IV criteria for current axis I disorders of major depression, panic disorder, obsessive-compulsive disorder, generalized anxiety disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder. The rationale for excluding them is that symptoms from these disorders may affect dependent variables and complicate interpretation of the data.
4. No use of benzodiazepines in excess of three times in the past two weeks by self report and urine drug screen.
5. Subjects must not be taking zolpidem (Ambien™), zaleplon (Sonata™), or eszopiclone (Lunesta™) in excess of three times in past two weeks.
6. No history of delirium tremens or alcohol withdrawal seizures.
7. Has current suicidal ideation with plan or homicidal ideation.
8. Need for maintenance or acute treatment with any psychoactive medication including antiseizure medications.
9. Use of disulfiram, naltrexone, acamprosate, or anticonvulsants in last 30 days.
10. Clinically significant medical problems such as cardiovascular, renal, GI, or endocrine problem that would impair participation or limit medication ingestion.
11. Sexually active females of child-bearing potential who are pregnant (by -beta HCG), nursing, or who are not using a reliable form of birth control.
12. Has current charges pending for a violent crime (not including DUI related offenses).
13. Has taken gabapentin or flumazenil in the last month or has experienced adverse effects from it at any time in the past.
14. Hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) greater than 3 times normal at screening.
15. Persons with metal implants or pacemaker since fMRI will be used.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC-Center for Drug and Alcohol Programs, Charleston, South Carolina, United States

REFERENCES:
- [Result] Anton RF, Myrick H, Baros AM, Latham PK, Randall PK, Wright TM, Stewart SH, Waid R, Malcolm R. Efficacy of a combination of flumazenil and gabapentin in the treatment of alcohol dependence: relationship to alcohol withdrawal symptoms. J Clin Psychopharmacol. 2009 Aug;29(4):334-42. doi: 10.1097/JCP.0b013e3181aba6a4. PMID 19593171
- [Result] Schacht JP, Randall PK, Waid LR, Baros AM, Latham PK, Wright TM, Myrick H, Anton RF. Neurocognitive performance, alcohol withdrawal, and effects of a combination of flumazenil and gabapentin in alcohol dependence. Alcohol Clin Exp Res. 2011 Nov;35(11):2030-8. doi: 10.1111/j.1530-0277.2011.01554.x. Epub 2011 Jun 1. PMID 21631542
- See also: Main Web Page for the MUSC-Center for Drug and Alcohol Programs — http://www.muschealth.com/cdap/

RESULTS

PARTICIPANT FLOW:
Groups:
- Low CIWA Flumazenil/Gabapentin; High CIWAar Flumazenil/Gabapentin: 2 mg flumazenil given over 20 minutes on Day 1 and Day 2. Gabapentin 300 mg Day 1; gabapentin 600 mg Day 2; gabapentin 900 mg Day 3; gabapentin 1200 mg Day 4 to 30; gabapentin 900 mg day 31-33; gabapentin 600 mg day 34-36; gabapentin 300 mg day 37-39.
- Low CIWAar Placebo; High CIWAar Placebo: 20 mg Saline infused slowly over 20 minutes. Placebo 1 capsule Day 1, 2 capsules Day 2, 3 capsules Day 3, 4 capsules days 4 to 30; 3 capsules Day 31 to 33; 2 capsules day 34 to 36 and 1 capsule 37 to 39.
Period: Overall Study
Arm/Group | Low CIWA Flumazenil/Gabapentin | Low CIWAar Placebo | High CIWAar Placebo | High CIWAar Flumazenil/Gabapentin
Started | 18 | 26 | 9 | 7
Completed | 18 | 26 | 9 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low CIWAar Placebo | Low CIWAar Flumazenil/Gabapentin | High CIWAar Placebo | High CIWAar Flumazenil/Gabapentin | Total
Number analyzed (Participants) | 18 | 26 | 9 | 7 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 26 | 9 | 7 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.2) | 44.1 (11.9) | 50.3 (8.5) | 46.7 (5.6) | 46.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 1 | 14
  Male | 14 | 20 | 6 | 6 | 46
Region of Enrollment [Number; unit: participants]
  United States | 18 | 26 | 9 | 7 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percent Subjects Completely Abstinent
Description: percent of subjects completely abstinent during the six week medication study study
Time Frame: 6 week trial
Measure: Number; unit: percent of participants
Arm/Group | Low CIWA Flumazenil/Gabapentin | Low CIWAar Placebo | High CIWAar Placebo | High CIWAar Flumazenil/Gabapentin
Number analyzed (Participants) | 18 | 26 | 9 | 7
percent of participants | 44 | 19 | 33 | 71
Statistical Analysis 1: Comparison: Low CIWA Flumazenil/Gabapentin vs Low CIWAar Placebo vs High CIWAar Placebo vs High CIWAar Flumazenil/Gabapentin; Test type: Superiority; p = 0.03, Regression, Logistic

2. Primary Outcome: Percent Days Abstinent
Description: percent days abstinent during treatment
Time Frame: Weeks 1 to 6
Measure: Mean (Standard Deviation); unit: percent days
Arm/Group | Low CIWA Flumazenil/Gabapentin | Low CIWAar Placebo | High CIWAar Placebo | High CIWAar Flumazenil/Gabapentin
Number analyzed (Participants) | 18 | 26 | 9 | 7
percent days | 70.8 (24.2) | 86.1 (20.7) | 75.9 (27) | 95.9 (9.7)
Statistical Analysis 1: Comparison: Low CIWA Flumazenil/Gabapentin vs Low CIWAar Placebo vs High CIWAar Placebo vs High CIWAar Flumazenil/Gabapentin; The analysis was an ANOVA interaction analysis with alcohol withdrawal (AW) group (Low vs. High) by medication group (active versus placebo medication) across the 6 weeks of the medication trial; Test type: Superiority; p = 0.0006, ANOVA — This p value is for the interaction of AW status by medication group

ADVERSE EVENTS:
Arm/Group | Low CIWA Flumazenil/Gabapentin | Low CIWAar Placebo | High CIWAar Placebo | High CIWAar Flumazenil/Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/26 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/18 | 0/26 | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No